CLINICAL TRIAL: NCT02556710
Title: A Randomized, Placebo-Controlled, Double-Blind Study to Evaluated the Efficacy and Safety of an Intra-Articular Injection of AMPION™ in Adults With Pain Due to Osteoarthritis of the Knee
Brief Title: A Study to Evaluate the Efficacy & Safety of an Intra-Articular Ampion Injection for Pain of Osteoarthritis of the Knee
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ampio Pharmaceuticals. Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AP-003-B
Record Dates: First submitted 2015-09-18; First posted 2015-09-22 (Estimated); Results first posted 2022-08-08 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: Osteoarthritis of the Knee
Keywords: Osteoarthritis; Osteoarthritis of the Knee
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AMPION™ 4 mL dose (Experimental): 4 mL injection of Ampion
  Interventions: Biological: 4 mL injection of AMPION™
- Placebo 4 mL dose (Placebo Comparator): 4 mL Injection of Placebo
  Interventions: Drug: 4 mL injection of Placebo

INTERVENTIONS:
Biological: 4 mL injection of AMPION™ — 4 mL Injection of Ampion
  Arms: AMPION™ 4 mL dose
Drug: 4 mL injection of Placebo — 4 mL Injection of Placebo
  Other Names: Saline
  Arms: Placebo 4 mL dose

SUMMARY:
This study will evaluate the efficacy and safety of an intra-articular injection of AMPION™ in adults with pain due to osteoarthritis of the knee

DETAILED DESCRIPTION:
A Randomized, Placebo-Controlled, Double-Blind Study To Evaluate The Efficacy And Safety Of An Intra-Articular Injection Of AMPION™ In Adults With Pain Due to Osteoarthritis Of The Knee

The primary trial objective is to evaluate the efficacy of 4 mL of AMPION™ versus 4 mL placebo intra-articular (IA) injection in improving knee pain, when applied to patients suffering from OA of the knee.

The secondary trial objective is evaluation of the safety of an intra-articular injection of AMPION™.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide written informed consent to participate in the study;
* Willing and able to comply with all study requirements and instructions of the site study staff;
* Male or female, 40 years to 85 years old (inclusive);
* Must be ambulatory;
* Index knee must be symptomatic for greater than 6 months with a clinical diagnosis of OA and supported by radiological evidence (Kellgren Lawrence Grade II, III, or IV) read by a central reader;
* WOMAC 5-point Likert pain subscale <1.5 in the contralateral knee;
* Moderate to moderately-severe OA pain in the index knee (rating of at least 1.5 on the WOMAC Index 3.1 5-point Likert Pain Subscale);
* Moderate to moderately-severe OA pain in the index knee (even if chronic doses of nonsteroidal anti-inflammatory drug (NSAID), which have not changed in the 4 weeks prior to screening, have been/are being used);
* Ability to discontinue NSAID use at Screening visit and/or 72 hours prior to the Baseline visit and for the duration of the clinical study (low dose Aspirin is allowed during the study);
* No analgesia (including acetaminophen [paracetamol]) taken 24 hours prior to an efficacy measure;
* No known clinically significant liver abnormality (e.g. cirrhosis, transplant, etc.).

Exclusion Criteria:

* As a result of medical review and screening investigation, the Principal Investigator considers the patient unfit for the study
* A history of allergic reactions to human albumin (reaction to non-human albumin such as egg albumin is not an exclusion criterion)
* A history of allergic reactions to excipients in 5% human albumin (N-acetyltryptophan, sodium caprylate)
* Presence of tense effusions
* Inflammatory or crystal arthropathies, acute fractures, history of aseptic necrosis or joint replacement in the affected knee, as assessed locally by the Principal Investigator
* Isolated patella femoral syndrome, also known as chondromalacia
* Any other disease or condition interfering with the free use and evaluation of the index knee for the duration of the trial (e.g. cancer, congenital defects, spine osteoarthritis)
* Major injury to the index knee within the 12 months prior to screening
* Severe hip osteoarthritis ipsilateral to the index knee
* Any pain that could interfere with the assessment of index knee pain (e.g. pain in any other part of the lower extremities, pain radiating to the knee)
* Any pharmacological or non-pharmacological treatment targeting OA started or changed during the 4 weeks prior to randomization or likely to be changed during the duration of the study
* Pregnancy or planning to become pregnant during the study.
* Use of the following medications:
* No IA injected pain medications in the study knee during the study
* No analgesics containing opioids.
* NSAIDs are not permitted during the study; acetaminophen is available as a rescue medication during the study from the provided supply.
* No topical treatment on osteoarthritis index knee during the study
* No significant anticoagulant therapy (e.g. Heparin or Lovenox) during the study (treatment such as low dose Aspirin and Plavix are allowed)
* No systemic treatments that may interfere with safety or efficacy assessments during the study
* No immunosuppressants
* No use of corticosteroids
* No human albumin treatment in the 3 months before randomization or throughout the duration of the study

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Howard Levy, MD, Study Director — Ampio Pharmaceuticals. Inc.
Locations (1):
- Ampio Pharmaceuticals, Englewood, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cole B, McGrath B, Salottolo K, Bar-Or D. LMWF-5A for the Treatment of Severe Osteoarthritis of the Knee: Integrated Analysis of Safety and Efficacy. Orthopedics. 2018 Jan 1;41(1):e77-e83. doi: 10.3928/01477447-20171114-05. Epub 2017 Nov 21. PMID 29156068

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects will be recruited from the population being seen by Investigators at the clinical sites participating in the study. In addition, notifications about the opportunity for subjects to participate in a clinical trial will be sent to referring physicians.
Pre-assignment Details: Ability to discontinue NSAID use at Screening visit and/or 72 hours prior to the Baseline visit and for the duration of the clinical study. No analgesia (including acetaminophen [paracetamol]) taken 24 hours prior to an efficacy measure.
Groups:
- 4 mL AMPION™: AMPION™: 4 mL Ampion Injection
- 4 mL Saline Placebo: Saline: 4 mL Saline Injection
Period: Overall Study
Arm/Group | 4 mL AMPION™ | 4 mL Saline Placebo
Started | 237 | 243
Completed | 226 | 237
Not Completed | 11 | 6
Not completed — Surgical treatment | 3 | 0
Not completed — Required proscribed pain medication | 2 | 1
Not completed — Lack of Efficacy | 1 | 0
Not completed — Worsening osteoarthritis | 1 | 0
Not completed — Moved out of state | 1 | 0
Not completed — Missing reason | 3 | 1
Not completed — Pain as lack of efficacy | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 4 mL AMPION™ | 4 mL Saline Placebo | Total
Number analyzed (Participants) | 237 | 243 | 480
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.6 (9.05) | 60.8 (8.84) | 61.2 (8.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 159 | 152 | 311
  Male | 78 | 91 | 169
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17 | 15 | 32
  Not Hispanic or Latino | 219 | 228 | 447
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 51 | 42 | 93
  White | 180 | 197 | 377
  More than one race | 3 | 3 | 6
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 237 | 243 | 480
Weight (kg) [Mean (Standard Deviation); unit: kg] | 91.49 (22.38) | 95.19 (22.32) | 93.36 (22.41)
BMI (kg/m^2) [Mean (Standard Deviation); unit: kg/m^2] | 32.94 (6.98) | 33.91 (7.58) | 33.43 (7.30)
Kellgren Lawrence Grade [Count of Participants; unit: Participants] — Kellgren-Lawrence grading is based on the radiologic features of osteoarthritis.
  Ann Rheum Dis. 1957;16:494-502.
  Grade II (Mild): Definite osteophytes, possible joint space narrowing.
  Grade III (Moderate): Moderate osteophytes, definite joint space narrowing, some sclerosis, possible bone-end deformity.
  Grade IV (Severe): Large osteophytes, marked joint space narrowing, severe sclerosis, definite bone-end deformity.
  Participants
    Kellgren-Lawrence Grade II | 50 | 51 | 101
    Kellgren-Lawrence Grade III | 122 | 125 | 247
    Kellgren-Lawrence Grade IV | 65 | 67 | 132
WOMAC Pain [Mean (Standard Deviation); unit: score on a scale] — The Western Ontario and McMaster Universities Arthritis Index (WOMAC) 3.1 evaluates Pain (5 items): during walking, using stairs, in bed, sitting or lying, and standing upright.
  Subjects respond to each subscale by using a 5-point Likert score. (0=none; 1=mild; 2=moderate; 3=severe; 4=extreme). Mean of the 5 scores constitutes the Baseline Pain Score. The minimum score on this scale is 0, and the maximum score is 4.
  Higher scores are indicative of higher levels of self-reported pain.
  score on a scale | 2.37 (0.56) | 2.33 (0.53) | 2.35 (0.54)
WOMAC Function [Mean (Standard Deviation); unit: score on a scale] — WOMAC 3.1 evaluates Physical Function (17 items): using stairs, rising from sitting, standing, bending, walking, getting in/out of a car, shopping, putting on/taking off socks, rising from bed, lying in bed, getting in/out of bath, sitting, getting on/off toilet, heavy/light domestic duties.
  Subjects respond to each by using a 5-point Likert score. (0=none; 1=mild; 2=moderate; 3=severe; 4=extreme). Mean of the 17 scores constitutes the Baseline Function Score. Minimum score is 0; maximum is 4.
  Higher scores indicate higher levels of limitations of self-reported physical function.
  score on a scale | 2.37 (0.64) | 2.34 (0.60) | 2.36 (0.62)

OUTCOME MEASURES:

1. Primary Outcome: Change in Knee Pain
Description: Mean Change in WOMAC A Pain (Western Ontario and McMaster Universities Arthritis Index) score from Baseline to 12 weeks. 5-point Likert scale (0=none to 4=extreme). A negative difference constitutes a decrease in pain with a greater negative value indicating a greater reduction in pain.
Time Frame: Scored at Baseline and 12 weeks
Population: Intent to Treat (ITT)
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | 4 mL AMPION™ | 4 mL Saline Placebo
Number analyzed (Participants) | 237 | 243
score on a scale | -0.91 [-1.03 to -0.80] | -0.89 [-1.01 to -0.77]
Statistical Analysis 1: Comparison: 4 mL AMPION™ vs 4 mL Saline Placebo; Test type: Superiority; p = 0.94, ANCOVA; Adjusted for baseline WOMAC Score

2. Secondary Outcome: Change in Knee Function
Description: Mean change in WOMAC C function score (Western Ontario and McMaster Universities Arthritis Index) from Baseline to 12 weeks. 5-point Likert scale indicating limitation of function (0=none to 4=extreme). A greater negative value indicates a improvement in function.
Time Frame: Scored at Baseline and 12 Weeks
Population: Per Protocol (PP)
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | 4 mL AMPION™ | 4 mL Saline Placebo
Number analyzed (Participants) | 213 | 222
score on a scale | -1.04 [-1.17 to -0.92] | -0.97 [-1.10 to -0.85]
Statistical Analysis 1: Comparison: 4 mL AMPION™ vs 4 mL Saline Placebo; Test type: Superiority; p = 0.53, ANCOVA; Adjusted for baseline WOMAC score

3. Post Hoc Outcome: Change in Knee Pain of Kellgren-Lawrence Grade IV Subset
Description: as for outcome 1
Time Frame: Scored at Baseline and 12 weeks
Population: KL Grade IV Subset of Intent to Treat (ITT)
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | AMPION™ 4 mL Dose | Placebo 4 mL Dose
Number analyzed (Participants) | 65 | 67
score on a scale | -0.81 [-1.02 to -0.61] | -0.62 [-0.85 to -0.40]
Statistical Analysis 1: Comparison: AMPION™ 4 mL Dose vs Placebo 4 mL Dose; Test type: Superiority; p = 0.35, ANCOVA — Adjusted for baseline WOMAC Score

ADVERSE EVENTS:
Time Frame: 12 Weeks
Description: Patients will be followed for the occurrence of Adverse Events until 12 weeks after the first dose of study medication.
Arm/Group | 4 mL AMPION™ | 4 mL Saline Placebo
All-Cause Mortality (participants affected / at risk) | 0/236 | 0/243
Serious Adverse Events (participants affected / at risk) | 2/236 | 4/243
Other Adverse Events (participants affected / at risk) | 47/236 | 44/243
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 4 mL AMPION™ (N=236) | 4 mL Saline Placebo (N=243)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cerebrovascular Accident (Nervous system disorders) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 0 (0) | 1 (1)
Malignant Melanoma In Situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Intussusception (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 4 mL AMPION™ (N=236) | 4 mL Saline Placebo (N=243)
Nasopharyngitis (Infections and infestations) | 10 (10) | 10 (10)
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 (11) | 8 (8)
Upper Respiratory Tract Infection (Infections and infestations) | 6 (6) | 13 (13)
Sinusitis (Infections and infestations) | 6 (6) | 4 (4)
Headache (Nervous system disorders) | 5 (5) | 2 (2)
Back Pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (2)
Hypertension (Vascular disorders) | 1 (1) | 4 (4)
Joint Swelling (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes